CLINICAL TRIAL: NCT04833335
Title: ASL in Diagnostics of Tumor Progression Versus Radionecrosis in Brain Metastasis Following Gamma Knife Treatment.
Brief Title: ASL in Brain Metastasis MRI Following Gamma Knife Treatment
Acronym: GK-ASL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190736
Record Dates: First submitted 2021-03-19; First posted 2021-04-06 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Brain Metastases
Keywords: ASL; MRI; Metastasis; Gamma knife; Radionecrosis
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with brain metastases treated with Gamma Knife whose lesions suggest tumor recurrence versus (Experimental): Inclusion visit, 1 month later, 6 month later
  Interventions: Other: MRI perfusion sequence

INTERVENTIONS:
Other: MRI perfusion sequence — Quantitative analysis
  Other Names: Arterial Spin Labeling (ASL)

SUMMARY:
Arterial spin labeling (ASL) is a non-invasive MRI technique that could help the radiologists to distinguish brain metastasis progression versus radionecrosis following gamma-knife treatment.

The primary target of the study is to establish the diagnostic performances (specificity, sensitivity) of quantitative measures of ASL in brain metastases suspected of progression/radionecrosis after GK treatment

DETAILED DESCRIPTION:
The metastasis progression versus radionecrosis following GK treatment can sometimes be difficult to distinguish. 60 patients will be included in this prospective, monocentric study. 3 MRI (baseline, 1month and 6 month follow-ups) will be performed. Two neuroradiologists will blindly analyse the MRIs comparing ASL sensibility and specificity to the standard morphological evaluation and T2 perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Brain metastasis from histologically proven tumor
* GK treatment within 4 month prior to the inclusion
* Lesions suspected of progression/ radionecrosis :

  i.e.≥ 25% of the size progression
* Lesion size: gadolinium enhanced part of the tumour ≥1 cm

Exclusion Criteria:

* Pregnancy
* Medical history of primitive brain tumour
* MRI incompatibility/ medical history of contrast agent allergy
* Claustrophobia
* Patient unable to consent
* Epilepsia/recent stroke
* Patients participating in other studies
* Patients without health care insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2028-09-24 (Estimated); Study Completion 2028-09-24 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of ASL quantitative analysis in brain metastasis following GK treatment : tumor perfusion with quantitative measurement (one value) of RCBF (relative cerebral blood flow) on the ASL sequence | Evolution between Baseline MRI, 1 and 6 month follow up MRI
  Quantitative analysis (rCBF) of the evolution of brain metastasis between the initiation of treatment and 6 months after.

SECONDARY OUTCOMES:
ASL Perfusion: Cerebral blood flow measurements | Baseline MRI, 1 and 6 month follow up MRI
Interreader correlation | Baseline MRI, 1 and 6 month follow-up MRI
  Two neuroradiologists
Morphological analysis of the lesions | Baseline MRI, 1 and 6 month follow-up MRI
  Lesion size, oedema

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neuroradiologie, hôpital Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No